CLINICAL TRIAL: NCT03362762
Title: Characteristics of Type 2 Diabetes Patients, Treated With Insulin and Their Follow up Care in Guadeloupe
Acronym: DT2IT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: RNI-PAP-913379
Record Dates: First submitted 2017-11-27; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Type 2 diabetes; insulin; Hb1Ac; glycemia; Guadeloupe
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Description of plans insuliniques used in Guadeloupe in the type 2 diabetes and the characteristics of the handled patients: — The physician or the endocrinologist will see the patient during his consultation. The pharmacist will see the patient when he goes to the pharmacy for an insulin treatment. In each case, the patient will be informed about the study, about the medical data that will be collected anonymously. The date will be strictly confidential and under medical secrecy. Then the patient will meet the physician during another consultation at the University Hospital Center of Guadeloupe, in order to collect information's on a questionnaire. Otherwise, the physician can meet the patient at his home, in case he can't move to the University Hospital Center of Guadeloupe.

SUMMARY:
Type 2 diabetes is a major problem of public health in the French West Indies, with an estimated prevalence of 8%, twice more than in France. In Guadeloupe, according to the statistical data of hospital morbidity in 2004, 2643 hospital stays were diagnosed with diabetes. These cases mainly concerned woman (62%) and the elderly, from 45 to 74 years old (67%).

The main objective of this research is to describe the insulin protocol used in Guadeloupe for treated type 2 diabetes patients and their characteristics:

* The duration of the type 2 diabetes
* Time elapsing between the diagnosis and the treatment by insulin
* Where the follow up care took place
* Existence of complications

Secondary objectives were to describe the link between the HbA1c rate and the insulin therapy protocol. And also to present the main inconveniences expressed by patients and their degree of autonomy.

DETAILED DESCRIPTION:
Nowadays the set up for insulin treatment is available in general practitioners' offices. However, it is restrained by the reticence of patients and physicians. For type 2 diabetes, insulin therapy is well managed and there is ongoing progress. But there are still some questions about the effect of the treatment in the everyday life of patients: culture, fear, material resources, necessity of education.

Ignorance and prejudices on insulin injection are still prevalent and often it delays for more than a year the time when patients have to switch an insulin treatment for unbalanced chronic disorder.

Type 2 diabetes patients think that the treatment is heavy, can lead to serious hypoglycemia, is uncomfortable for family and can cause fear.

Education of the patients can reduce ignorance and prejudices about insulin treatment.

Nowadays studies show that diabetes patients want to be more involved in the decisions linked to their treatment which impact their perception of the disease and the treatment.

Auto measurement of glycaemia can help the patient better manage his disease and make him understand the importance of controlling his glycaemia levels.

This study could allow to:

* Offer a new care organization for a better use of resources (network, patient therapeutic education…)
* Set up adequate training for professionals and for patients being cared for in medical offices.
* Improve the glycemic balance of patients and slower the growth of degenerative complications.

ELIGIBILITY:
Inclusion Criteria:

* Men or woman
* Age ≥ 18 years old
* Patient with type 2 diabetes, treated with insulin for at least one year
* Patient accepting to participate to the study

Exclusion Criteria:

• Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns the type 2 diabetes patients, followed by physicians in Guadeloupe.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2016-09-27 (Actual)

PRIMARY OUTCOMES:
Characteristic of type 2 diabetes patients, treated with insulin in Guadeloupe | Trough study completion, an average of 2 years
  A descriptive analysis will be done on the population concerned by the study, for the socio demographic, clinical and therapeutic characteristics.
  * the duration of the type 2 diabetes,
  * time elapsing between the diagnostic and the treatment by insulin,
  * place of the follow up care,
  * existence of complications.

SECONDARY OUTCOMES:
Describe the relation between the rate of HbAC and the plan of insulinothérapie | Trough study completion, an average of 2 years
  Sreening of HbAC

CONTACTS AND LOCATIONS:
Overall Officials: Pauline NOUVIER KANGAMBEGA, medicine degree, diabetes, Principal Investigator — Hospital University Center of Pointe-à-Pitre
Locations (1):
- University Hospital Center of Pointe-à-Pitre, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No